CLINICAL TRIAL: NCT04597034
Title: A Randomized, Controlled Trial to Evaluate Efficacy and Safety of a Highly Selective Semipermeable Membrane (AN-69 Oxiris) in Comparison With a Semi Selective Semipermeable Membrane (Standard AN-69) in COVID-19 Associated Acute Kidney Injury: oXAKI-COV Study.
Brief Title: Efficacy and Safety of a Highly Selective Semipermeable Membrane (AN-69 Oxiris) vs (Standard AN-69) in COVID-19
Acronym: oXAKI-COV
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Instituto Nacional de Ciencias Medicas y Nutricion Salvador Zubiran (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NMM-3401-20-20-1
Record Dates: First submitted 2020-10-03; First posted 2020-10-22 (Actual); Last update posted 2020-10-22 (Actual); Status verified 2020-09

CONDITIONS: Covid19; AKI
Keywords: COVID-19; AKI; CRRT; AN69 Oxiris; AN69 Standar
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Intervention Model Description: Randomized,open-label, controlled trial in critically ill patients with suspected or confirmed COVID-19 disease, AKI, and criteria for continuous renal replacement therapy initiation admitted in any of the two participating institutions. Patients meeting inclusion criteria will be randomized to receive CRRT with AN69-Oxiris membrane or standard AN69 membrane during a 72h period.
Who Masked: Participant
Masking Description: Group allocation for the AN-69 Oxiris membrane or the standard AN-69 membrane will be done by randomization before starting each CRRT treatment. This process will be performed through Epidat 4.2 software by one of the researchers from the Instituto Nacional de Ciencias Médicas y Nutrición, Salvador Zubirán.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- AN69 Oxiris (Experimental): * To evaluate the safety in using the AN69-Oxiris membrane in contrast with the use of a conventional membrane in critically ill patients with COVID-19 associated AKI and CRRT requirements.
  * To examine the efficacy of the AN69-Oxiris membrane in reducing inflammatory interleukins compared with reduction using conventional membranes in this specific group of patients.
  * To exhibit the potential benefit of AN69-Oxiris in decreasing ICU length of stay versus the effect of using conventional membranes in COVID-19 associated AKI.
  * To investigate the effect of AN69-Oxiris in reducing 28-day mortality in contrast compared with the effect of a conventional membrane in this population.
  Interventions: Procedure: AN69-Oxiris
- AN69 Standard (Active Comparator): * To evaluate the safety in using the AN69-Oxiris membrane in contrast with the use of a conventional membrane in critically ill patients with COVID-19 associated AKI and CRRT requirements.
  * To examine the efficacy of the AN69-Oxiris membrane in reducing inflammatory interleukins compared with reduction using conventional membranes in this specific group of patients.
  * To exhibit the potential benefit of AN69-Oxiris in decreasing ICU length of stay versus the effect of using conventional membranes in COVID-19 associated AKI.
  * To investigate the effect of AN69-Oxiris in reducing 28-day mortality in contrast compared with the effect of a conventional membrane in this population.
  Interventions: Procedure: AN69-Standard

INTERVENTIONS:
Procedure: AN69-Oxiris — To demonstrate clinical efficacy of AN69-Oxiris membrane to reach a stable MAP, with less vasopressor dosing (at least 0.1 micrograms/kg/min) after 72h of treatment, compared to a conventional membrane (standard AN69) in critically ill patients with AKI, COVID-19 infection and requirement of continuous renal replacement therapy.
  Arms: AN69 Oxiris
Procedure: AN69-Standard — Standard treatment.
  Arms: AN69 Standard

SUMMARY:
Abstract Title: Randomized,open-label, controlled trial to evaluate efficacy and safety of a highly selective semipermeable membrane (AN69-Oxiris) in comparison with a selective semipermeable membrane ( standard AN69) in COVID-19 associated acute kidney injury: oXAKI-COV study Rationale: Acute kidney injury (AKI) in critically ill mechanically ventilated patients with COVID-19 disease, is present in up to 30% of this group and more than 50% of them will need renal replacement therapy in the form of continuous renal replacement therapy (CRRT). Acute kidney injury in this context seems to be a marker of multiorgan dysfunction and it produces increased mortality in this population. There is a vast amount of mechanisms that lead to AKI in critically ill patients with COVID-19; however, the cytokine storm could be the strongest mechanism implicated in AKI development in individuals with continuous renal replacement therapy requirements. Therefore, blocking or reducing the cytokine storm is thought to be a therapeutic target.

Highly selective semipermeable membranes (AN69-Oxiris) have been shown able to adsorb endotoxins and to eliminate inflammatory cytokines, thus representing a valuable therapeutic option in this infection.

Objective: To demonstrate clinical efficacy of AN69-Oxiris membrane to reach a stable MAP, with less vasopressor dosing (at least 0.1 micrograms/kg/min) after 72h of treatment, compared to a conventional membrane (standard AN69) in critically ill patients with AKI, COVID-19 infection and requirement of continuous renal replacement therapy.

Study design: Randomized,open-label, controlled trial in critically ill patients with suspected or confirmed COVID-19 disease, AKI, and criteria for continuous renal replacement therapy initiation admitted in any of the two participating institutions. Patients meeting inclusion criteria will be randomized to receive CRRT with AN69-Oxiris membrane or standard AN69 membrane during a 72h period.

DETAILED DESCRIPTION:
On March 11th, 2020 the World Health Organization declared the new coronavirus disease (COVID-19) as a global pandemic. In México, approximately 35% of COVID-19 positive patients require hospital admission and 4.4% do it in the intensive care unit. Acute kidney injury (AKI) in mild to moderate COVID-19 disease seems to be infrequent; in contrast, critically ill patients or those with a severe disease develop AKI in up to 30% of the cases and nearly half of them will need renal replacement therapy in the form of continuous renal replacement therapy (CRRT). AKI in this context seems to be a marker of multiorgan dysfunction and it produces increased mortality in this population.

Multiple mechanisms of AKI in COVID-19 disease have been proposed: direct injury into podocytes and proximal convoluted tubule cells, organ-organ interactions (lung-kidney axis), and cytokine storm. Of them, the severe cytokine-induced injury seems to be the strongest mechanism participating in AKI in this group of severely ill patients with CRRT need thus representing a valuable therapeutic option.

Lately, extracorporeal blood purification therapies have been proposed as a therapeutic tool for cytokine removal in patients with sepsis (prototype of cytokine storm model). Therefore, new membranes with hemoadsorption capacity have been developed and are now commercially available. The first group of membranes used for patients with sepsis and inflammatory systemic response syndrome was high cut-off semipermeable membranes (HCO) followed by non-selective adsorbent membranes, semi selective semipermeable membranes (AN69), and last highly selective semipermeable (especially those with endotoxin and cytokine adsorption, such as AN69-Oxiris). Although these membranes were designed to improve inflammation, they can also be used as a regular filter in CRTT in patients with AKI. These products can be purchased in our country and internationally but there is scant evidence supporting its efficacy to improve clinical outcomes in patients with overt sepsis.

Highly selective semipermeable membranes (AN69-Oxiris) possess a great capacity for endotoxin adsorption and cytokine removal (interleukin 6 [IL-6], tumor necrosis factor-alfa [TNF-α], C reactive protein [CRP] , and interleukin 1b), representing a valuable therapeutic option in septic shock; these findings have been tested mainly in experimental models. There are human-based studies with non-representative statistical samples in which these membranes appear to improve severity scores without any impact in mortality. This membrane has been used in some regions around the world during the COVID-19 pandemic; recently, Ma et al published two severe COVID-19 patients who were treated with AN69-Oxiris resulting in decreased levels of inflammatory markers (ie, CRP and IL-6) and better lymphocyte counts. However, there is uncertainty in the clinical benefit of those changes.

Given the lack of specific drugs or vaccine targeted for COVID-19 and, taking into account the pathophysiologic basis that supports the use of extracorporeal blood purification therapies to reduce the cytokine storm in COVID-19 infected patients with AKI requiring CRRT, the use of these membranes could be of clinical utility in the disease. Here our group presents a randomized,open-label, controlled trial to evaluate efficacy and safety of a highly selective semipermeable membrane (AN69-Oxiris) in comparison with a semi selective semipermeable membrane ( standard AN69) in COVID-19 associated acute kidney injury.

Hypothesis Research question: In critically ill patients with COVID-19 disease and AKI requiring CRRT, is the AN69-Oxiris membrane of greater benefit to sustain MAP a lower vasopressor dose in comparison with a conventional AN69 standard membrane, after 72 hours of treatment?

Alternative hypothesis: The use of the AN69-Oxiris membrane will decrease vasopressor requirement in at least 0.1 micrograms/kilogram/minute to sustain a stable MAP in contrast with the usage of AN69 standard membrane, in critically ill patients with COVID-19 and AKI requiring CRRT after 72 h of treatment.

Goals Primary goal: To demonstrate the clinical efficacy of AN69-Oxiris in decreasing vasopressor requirement in at least 0.1 micrograms/kilogram/minute to sustain a stable MAP in contrast with the usage of AN69 standard membrane, in critically ill patients with COVID-19 and AKI requiring CRRT after 72 h of treatment.

Exploratory goals:

* To evaluate the safety in using the AN69-Oxiris membrane in contrast with the use of a conventional membrane in critically ill patients with COVID-19 associated AKI and CRRT requirements.
* To examine the efficacy of the AN69-Oxiris membrane in reducing inflammatory interleukins compared with reduction using conventional membranes in this specific group of patients.
* To exhibit the potential benefit of AN69-Oxiris in decreasing ICU length of stay versus the effect of using conventional membranes in COVID-19 associated AKI.
* To investigate the effect of AN69-Oxiris in reducing 28-day mortality in contrast compared with the effect of a conventional membrane in this population.

ELIGIBILITY:
Inclusion Criteria:

1. Patients aged ≥ 18 years old.
2. A diagnosis of a confirmed, defined by a positive rt-PCR for SARS CoV-2, or suspected COVID-19 disease, with suggestive findings on a chest CT scan.
3. Patients on mechanical ventilation.
4. The presence of an informed consent signed by the next of kin.
5. Patients with KDIGO AKI stage 2: defined by a rise in creatinine 2-2.9 times baseline and/or a urinary output less than 0.5 ml/kg/hr for 12 hours, with failure after a furosemide stress test.
6. The use of vasopressor, any dose.
7. Complete medical history and complete laboratories.

Exclusion Criteria:

1. Chronic kidney disease KDIGO stage 4, 5, or 5D.
2. Next of kin unwilling or patient unwilling to participate.
3. Patients with a life expectancy of fewer than 72 hours according to the attending physician criteria.
4. Patients older than 75 years.
5. Patients with SOFA > 11.
6. Patients with severe liver failure.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Estimated)
Dates: Start 2020-10-02 (Actual); Primary Completion 2021-12-30 (Estimated); Study Completion 2022-03-30 (Estimated)

PRIMARY OUTCOMES:
Primary outcome: | 90 days
  Change in norepinephrine requirement by at least 0.1 micrograms / kg / min to maintain similar MAP after initiation of CRRT with Oxiris membrane compared to standard AN69 membrane. MAP measurements will be performed hourly and norepinephrine requirement will be recorded at that time.

SECONDARY OUTCOMES:
Secondary outcomes measures: | 72 hours
  Effectiveness of the AN69-Oxiris membrane in reducing interleukin serum levels (IL 6, IL 10, and TNF alpha).
  Serum will be taken every 8 hours for its measurement by ELISA method.
Secondary outcomes measures: | 30 days
  To establish the safety (the same risk infection and bleeding) of using the AN69- Oxiris membrane in patients with AKI and COVID-19 infection who require CRRT.
  Gross bleeding events (gastrointestinal or urinary) as well as catheter-associated infection events (criteria according to IDSA) will be recorded.
Secondary outcomes measures: | 90 days
  Length of stay in UCI among patients who used AN69-Oxiris membrane in compared to the use of a conventional membrane (standard AN-69) in critically ill patients with COVID-19 associated AKI and CRRT requirement.

CONTACTS AND LOCATIONS:
Locations (1):
- Instituto Nacional de Ciencias Médicas y Nutrición Salvador Zubirán, Mexico City, Mexico

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Ronco C, Reis T. Kidney involvement in COVID-19 and rationale for extracorporeal therapies. Nat Rev Nephrol. 2020 Jun;16(6):308-310. doi: 10.1038/s41581-020-0284-7. PMID 32273593
- [Result] Ronco C, Reis T, De Rosa S. Coronavirus Epidemic and Extracorporeal Therapies in Intensive Care: si vis pacem para bellum. Blood Purif. 2020;49(3):255-258. doi: 10.1159/000507039. Epub 2020 Mar 13. No abstract available. PMID 32172242
- [Result] RENAL Replacement Therapy Study Investigators; Bellomo R, Cass A, Cole L, Finfer S, Gallagher M, Lo S, McArthur C, McGuinness S, Myburgh J, Norton R, Scheinkestel C, Su S. Intensity of continuous renal-replacement therapy in critically ill patients. N Engl J Med. 2009 Oct 22;361(17):1627-38. doi: 10.1056/NEJMoa0902413. PMID 19846848
- [Result] Morgera S, Haase M, Kuss T, Vargas-Hein O, Zuckermann-Becker H, Melzer C, Krieg H, Wegner B, Bellomo R, Neumayer HH. Pilot study on the effects of high cutoff hemofiltration on the need for norepinephrine in septic patients with acute renal failure. Crit Care Med. 2006 Aug;34(8):2099-104. doi: 10.1097/01.CCM.0000229147.50592.F9. PMID 16763508

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2020-10-17): https://cdn.clinicaltrials.gov/large-docs/34/NCT04597034/Prot_SAP_ICF_000.pdf